CLINICAL TRIAL: NCT04864457
Title: Alterations in the Transcription, Metabolism and Gut Microbiome in Young Adults With Coronary Syndrome Severity
Brief Title: Multi-omics Study of Young Adults Coronary Syndrome Patients
Acronym: Young-COSMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Young-COSMOS.001
Record Dates: First submitted 2020-11-29; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cell, plasma, faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal: Patients without coronary atherosclerotic burden
- Chronic coronary syndrome (CCS): CCS covers the different stages of development of coronary heart disease in addition to the clinical manifestations dominated by acute coronary thrombosis, including asymptomatic myocardial ischemia, vasospasm, and microcirculatory lesions. The six most common types of CCS include:Suspected coronary heart disease and "stable" angina symptoms, whether or not patients with dyspnea; Patients with newly emerged heart failure or left ventricular dysfunction suspected of CAD; Patients with no symptoms or stable symptoms within 1 year after ACS, or patients with recent revascularisation; Patients with or without symptoms more than 1 year after initial diagnosis or revascularization; Patients with angina pectoris, suspected vasospasm or microcirculatory diseases; Asymptomatic patients with coronary heart disease are found during screening.
- Acute coronary syndrome (ACS): ACS is a group of clinical syndromes commonly characterized by acute myocardial ischemia, including unstable angina pectoris (UA); Acute non-ST-segment elevation myocardial infarction (NSTEMI); Acute ST-segment elevation myocardial infarction (STEMI).

SUMMARY:
With the rapid development of China's economy, changes in diet structure, lifestyle and excessive mental pressure have led to a younger trend in the incidence of ACUTE coronary syndrome, and the mortality rate has been on the rise, especially in Shenzhen, the country with the youngest average age.Coronary heart disease among young people not only reduces the quality of life and loses the ability to work, but also prematurely consumes medical resources and increases social costs, bringing heavy burdens to families and society.Therefore, it is of great significance to conduct researches on the transcription, metabolism and microbiome of young patients with ACUTE coronary syndrome and obtain the multi-group characteristics of these patients for early warning, guiding the improvement of life style, regulating treatment, improving treatment rate, and reducing family and social burden.

DETAILED DESCRIPTION:
1. Research purpose and significance In recent years, with the rapid development of China's economy, the changes in dietary structure and lifestyle, as well as excessive mental stress, and other factors have led to an obvious trend of younger incidence of Coronary artery disease (CAD), and an increase in the death rate.This is especially true in Shenzhen, which has the youngest average age in the country.CAD in young people not only reduces the quality of life and loses the ability to work, but also prematurely consumes medical resources, increases social costs, and brings heavy burden to families and society.Therefore, it is of great significance to study the transcriptome, metabolome and intestinal flora of young CAD and obtain the multiomic characteristics of these patients for early warning, guiding the improvement of lifestyle, regulating treatment, improving treatment rate, and reducing the burden of family and society.

2. Research status at home and abroad

1. The public health burden of coronary artery disease in China With the development of social economy, China's national lifestyle has undergone profound changes. Under the social background of population aging and urbanization, the risk of Atherosclerotic cardiovascular disease (ASCVD) is increasing day by day.The incidence of cardiovascular diseases continues to increase.ASCVD is the number one cause of death in China, surpassing cancer and other diseases.CAD is an important part of ASCVD. According to China Cardiovascular Health and Disease Report 2019, the total number of CAD patients in China is about 11 million.CAD causes extremely high mortality and disability rate, causing serious public health burden and social and economic burden.The 5th Chinese health service survey in 2013 showed that the prevalence rate of coronary artery disease among residents ≥15 years old was 12.3‰ in urban areas, 8.1‰ in rural areas, and 10.2‰ in urban and rural areas.According to China's Health Statistics Yearbook 2018, the mortality rate from coronary artery disease was 115.32 per 100,000 urban residents and 122.04/100,000 rural residents in 2017.Based on the sample database of inpatients insured by China's basic medical insurance from 2010 to 2014, the annual hospitalization rate of acute myocardial infarction was estimated to be 44.2/100,000.The median hospitalization cost for patients with acute myocardial infarction in urban China is 31,000 yuan, and the median hospitalization cost for patients receiving coronary intervention therapy is 52,000 yuan.

   It is an indisputting fact that CAD causes serious social burden. How to let more CAD patients find their disease as early as possible, intervene as early as possible, and avoid returning to poverty, becoming disabled or even dying due to disease due to the aggravation of disease is an urgent public health problem.According to the Healthy China 2030 Plan, the premature mortality rate from major chronic diseases is expected to drop from 18.5% in 2015 to 15.9%, indicating that the management of chronic diseases is also being increasingly emphasized at the national health policy-making level.
2. Epidemiological characteristics of coronary heart disease in young people With the improvement of diagnosis and treatment level and people's attention to CAD, the case fatality rate of CAD in the world has decreased significantly.Epidemiological data in the United States showed that from 1980 to 2002, the mortality rate of male and female CAD patients decreased by 52% and 49% respectively [3].Unfortunately, improvements in CAD outcomes have not covered all age groups.Epidemiological data from the United States [3], the United Kingdom [4], Canada [5] and Australia [6] all show that the morbidity and mortality of young CAD patients younger than 45 years old are increasing year by year.The research group also confirmed in the previous study that the proportion of young CAD patients admitted to the Department of Cardiology of Shenzhen People's Hospital increased year by year from 2015 to 2019.This shows that young CAD patients have different disease development characteristics, and the theory and basis of young CAD are derived from the study of the whole population, and the corresponding innovation of treatment concept has not significantly improved the prognosis of young CAD patients.Therefore, it is of great significance to promote the research of youth CAD, reveal the pathogenesis of youth CAD, and explore the prediction, diagnostic markers and therapeutic targets for the prevention and treatment of youth CAD and the improvement of national health level.

   Compared with the general population, young CAD patients are often associated with multiple risk factors.According to statistics, more than half of the young people aged 18-24 have at least one CAD risk factor [9, 10], and nearly 1/4 of the young people have atherosclerotic plaques. The size and range of atherosclerotic plaques are directly positively correlated with the number of risk factors.Poor diet, overweight, hyperlipidemia, physical inactivity, and smoking are the major risk factors for young adults, and the number of risk factors is closely related to long-term outcomes.Ignorance of relevant risk factors in young people further increases the risk of CAD, and once coronary atherosclerotic plaque forms, the condition continues to progress to coronary artery disease, which will seriously affect the quality of life and life expectancy of young patients [11-13].However, at present, there are very few researches on the mechanism behind the special epidemiological phenomenon of CAD in young people [7, 8], and corresponding researches are urgently needed to explain the pathogenesis of this unique CAD population.
3. Dynamic pathological changes of coronary artery disease CAD is a chronically progressive, dynamically changing pathological process that can be in a long-term stable state or become unstable at any time. Plaque rupture or erosion can cause acute thrombotic events.According to clinical manifestations, CAD can be divided into Acute coronary syndrome (ACS) and Chronic coronary syndrome (CCS).

   ACS is a group of clinical syndromes characterized by acute myocardial ischemia, including ① unstable angina pectoris (UA);② Acute non-ST segment elevation myocardial infarction (NSTEMI);③ Acute ST-segment elevation myocardial infarction (STEMI).The main mechanism is the rupture or erosion of coronary atherosclerotic plaque combined with thrombosis and/or vasospasm, which causes the sharp aggravation of coronary artery stenosis or acute occlusion.

   CCS covers the different developmental stages of CHD in addition to the clinical manifestations dominated by acute coronary thrombosis, including asymptomatic myocardial ischemia, vasospasm, and microcirculatory lesions.The six most common CCS clinical conditions include: (1) patients with suspected coronary heart disease and "stable" angina pectoris, with or without dyspnea;② patients with newly emerged heart failure or left ventricular dysfunction, suspected of CAD;③ Patients with asymptomatic or stable symptoms within 1 year after ACS, or patients with recent revascularization;(4) Patients with or without symptoms at least 1 year after initial diagnosis or revascularization;⑤ patients with angina pectoris, suspected vasospasm or microcirculation diseases;(6) Asymptomatic patients with coronary heart disease were found during screening.

   The dynamic pathological process of CAD has become the focus of current research, and every link in the pathophysiological process may become a potential new target for prevention and treatment.
4. Research status of transcription, metabolism and intestinal flora of coronary artery disease Recent studies have shown that CAD is associated with changes in intestinal microbiota in different populations, and metabolites of intestinal microbiota are considered to be major markers of heart damage.Koren et al. found that the atherosclerotic plaques contained DNA sequences of bacteria such as Staphylococcus aureus, Veroncoccus and Streptococcus, which could also be observed in the plaques of the intestinal vessels of the same individual.Liu et al. conducted multi-omics analysis on 161 CAD patients and 40 healthy controls, and found that the composition of intestinal flora and metabolites significantly changed with the severity of CAD.These studies suggest that intestinal flora can influence the dynamic pathological process of CAD by regulating the metabolic pathways of the host.

   Some special non-coding RNA molecules, such as circRNAs (Circularrnas) and Long non-coding RNAs (lncRNAs), were abnormally expressed during the development of CAD and had certain regulatory functions.As a biomarker and therapeutic target, it plays an important role in the diagnosis and treatment of CAD.At the same time, previous transcriptome analysis of a variety of atherosclerotic cells, animal and human vascular tissues revealed that a large number of genes were expressed abnormally during the pathological process of CAD [1-7], suggesting that these genes may be involved in the pathological process of CAD, but whether these genes are susceptible genes for young CAD remains unclear.
5. Our project ideas CAD in young people imposes a heavy burden on families and society.Young CAD has its own characteristics of the disease, and the elderly patients are different, smoking, drinking, staying up late and other bad lifestyle, as well as unreasonable diet, work pressure is more common in young CAD patients.Previous omics studies on CAD were conducted in the whole population and could not accurately reveal the pathogenesis of the young population.Therefore, only by studying the transcriptome, intestinal flora and metabolism of young CAD, revealing its pathogenesis and exploring new biomarkers and therapeutic targets, can we fundamentally solve the problems of young CAD and provide effective strategies for clinical prevention and treatment of young CAD.

This topic proposed line selected 18 to 45 years old coronary interventional diagnosis and treatment of 200 patients, according to the results of coronary angiography and clinical manifestations of divided into young patients with normal coronary group (40 cases), the young patients with chronic coronary syndrome group (80 cases) and youth group (80 cases), acute coronary syndrome patients to metabolism of the full spectrum of blood group and the whole transcriptome sequencing,And intestinal microflora metagenome and full spectrum metabolome sequencing of feces.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of normal coronary artery, chronic coronary syndrome or acute coronary syndrome by coronary angiography and clinical symptoms
* 18-45 years old

Exclusion Criteria:

* Patients with gastrointestinal diseases, recent 3 months of diarrhea, malignant tumors, autoimmune diseases and infectious diseases
* Patients with renal insufficiency (severe kidney disease creatinine > 267 mol/L)
* Patients with gastrointestinal surgery history within 1 year
* Patients with antibiotic use for more than 3 days within 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18 to 45 years with normal coronary artery, chronic coronary syndrome or acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Frequencies of alteration of RNA expression | During sample collection (1 year)
  The alteration of RNA expression, including mRNA, circRNA, and lncRNA, will be compared among young patients with normal coronary artery, chronic coronary syndrome and acute coronary syndrome by transcriptome sequencing.
Frequencies of alteration of gut microbiome | During sample collection (1 year)
  The alteration of Gut Microbiome will be compared young patients with normal coronary artery, chronic coronary syndrome and acute coronary syndrome by metagenomic tests on fecal DNA with the Illumina NovaseQ6000 sequencing platform.

SECONDARY OUTCOMES:
Alteration of inflammatory factors | During sample collection (1 year)
  The alteration of inflammatory factors, including hCRP, IL-8, IL-1b, IL-10 and TNF-a, will be compared among young patients with normal coronary artery, chronic coronary syndrome and acute coronary syndrome by ELISA
Alteration of dietary habit | During sample collection (1 year)
  The alteration of the dietary habit will be compared among young patients with normal coronary artery, chronic coronary syndrome and acute coronary syndrome by Eating Behaviors Questionnaire.
Frequencies of alteration of metabolites | During sample collection (1 year)
  The alteration of metabolites will be compared among young patients with normal coronary artery, chronic coronary syndrome and acute coronary syndrome by untargeted metabonomics assay based on LC/MS with Thermo Q ExactiveTM HF(X)

CONTACTS AND LOCATIONS:
Overall Officials: Shaohong Dong, MD, Study Chair — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China